CLINICAL TRIAL: NCT06578689
Title: Factors and Consequences Associated With Diabetic Foot Problems Among Diabetic Patients in Jordan
Status: Recruiting | Type: Observational
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Principal Investigator, Samah Al-Shatnawi, Associate Professor, King Abdullah University Hospital
Other Study IDs: 20240097
Record Dates: First submitted 2024-08-19; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM with DFU
  Interventions: Behavioral: Education
- DM without DFU

INTERVENTIONS:
Behavioral: Education — The control group received standard care, while the intervention group received standard care supplemented with formal educational session followed by ongoing education on foot care using mobile health by a clinical pharmacist.
  Groups: DM with DFU

SUMMARY:
Purpose: To assess diabetic foot ulcers (DFU)-related risk factors and complications among diabetes mellitus (DM) patients in Northern Jordan. Also, to analyze the impact of educational intervention on their behavior.

Methods: The study consisted of two phases. Phase one was a prospective cross-sectional study of 200 DM patients, including 94 with a history of DFU, where demographic and clinical data were collected to assess diabetic foot-associated risk factors and complications. Phase two was a randomized clinical trial with 105 DM patients: 52 in the control group received standard care, while 53 in the intervention group received standard care supplemented with formal educational session and ongoing foot care education via mobile health by a clinical pharmacist. Foot care practices and medication adherence were evaluated at baseline and after 8 weeks of follow-up.

DETAILED DESCRIPTION:
Background: Diabetes mellitus (DM) is a common chronic metabolic condition with numerous consequences, including diabetic foot ulcers. diabetic foot ulcer (DFU) is the major cause of non-traumatic lower extremity amputations. DFU is linked to several risk factors, including a lack of information and inadequate foot care practices. In Jordan, statistics on diabetic foot are few, with no evidence of the impact of patient education on disease outcomes.

Aims: To assess DFU-related risk factors and complications among DM patients in Northern Jordan. Also, analyze the impact of educational intervention on their behavior.

Methods: A prospective cross-sectional sample of 200 DM patients, including 94 with a history of DFU was initially selected. Subsequently, a smaller cohort of 105 patients was randomized into either a control group or an intervention group after providing written informed consent. The control group received standard care, while the intervention group received standard care supplemented with formal educational session followed by ongoing education on foot care using mobile health by a clinical pharmacist. Diabetic foot-associated risk factors and complications were assessed. Foot care practices and medication adherence were evaluated for both the control and intervention groups at baseline and again after 8 weeks of follow-up. Binary logistic regression was employed to assess factors associated with DFU. The Chi-square test and independent sample t-test were used to compare the behavior between the two groups before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults DM (1 year)

Have a mobile phone

Exclusion Criteria:

* Cognitive impairment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DM patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of diabetic patients without diabetic foot ulcers | 8 weeks
  Patients diagnosed with DM and have no reported DFU
Number of patients with diabetic foot ulcers | 8 weeks
  Patients diagnosed with DM and have been diagnosed with DFU
Number of patients receiving diabetic foot care education | 8 weeks
  Patients diagnosed with DM and received diabetic foot care education

SECONDARY OUTCOMES:
Number of patients reporting good foot care practices | 8 weeks
  Patients diagnosed with DM and DFU
Number of patients reporting Medication adherence | 8 weeks
  Patients diagnosed with DM and DFU

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Data was collected anonyms and coded